CLINICAL TRIAL: NCT06691217
Title: Effects of IL-1 Beta Inhibition on Vascular Inflammation in TET2 Clonal Hematopoiesis
Acronym: TECTONIC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Broad Institute of MIT and Harvard (Other); Yale University (Other)
Responsible Party: Principal Investigator, Michael C. Honigberg, MD, MPP, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024P002825
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Vascular Inflammation; ASCVD; ASCVD Management
Keywords: CHIP; TET2 CHIP; Clonal Hematopoiesis; Vascular Inflammation; ASCVD; ASCVD management
MeSH Terms: interventions — canakinumab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized, double-blind clinical trial of individuals with established coronary heart disease.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo: Control (Placebo Comparator): Participants with and without TET2 CHIP will receive placebo injection every 3 months for 4 doses as part of the randomized clinical trial part of this proposal.
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)
- Treatment: Canakinumab (Experimental): Participants with and without TET2 CHIP will receive 150mg of canakinumab every 3 months for 4 doses as part of the randomized clinical trial part of this proposal.
  Interventions: Drug: CANAKINUMAB (ILARIS®)

INTERVENTIONS:
Drug: CANAKINUMAB (ILARIS®) — Participants with and without TET2 CHIP will receive 150mg of canakinumab every 3 months for 4 doses as part of the randomized clinical trial part of this proposal.
  Arms: Treatment: Canakinumab
Drug: Saline (NaCl 0,9 %) (placebo) — Participants with and without TET2 CHIP will receive placebo injection every 3 months for 4 doses as part of the randomized clinical trial part of this proposal.
  Arms: Placebo: Control

SUMMARY:
The primary goal of this clinical trial is to test the hypothesis that the drug canakinumab (anti-IL-1B monoclonal antibody) decreases vascular inflammation when used by people with a history of coronary artery disease, including those with and without clonal hematopoiesis driven by mutations in TET2.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled study to test the effects of canakinumab, an inhibitor of interleukin-1B, on vascular inflammation in individuals with coronary artery disease. Half of the trial population will have clonal hematopoiesis of indeterminate potential (CHIP) driven by mutations in TET2. Participants (total N=120) will be randomized 1:1 to receive canakinumab (n=60) versus placebo (n=60). Baseline assessment in all participants will include coronary CT angiography, and a subset of participants in each group (n=16 per group) will undergo SPECT imaging to assess macrophage-specific vascular inflammation. After randomization, participants will have injection/safety visits at Week 0, Week 12, Week 24, and Week 36. Repeat imaging assessments for vascular inflammation will occur during the Week 48 visit(s). Participants will undergo final study and safety assessments at Week 60. The primary endpoint is change in the fat attenuation index (FAI) as measured by coronary CT angiography between baseline and Week 48. Other key endpoints are change in macrophage-specific inflammation by SPECT between baseline and Week 48 and change in TET2 clonal variant allele fraction among participant with TET2 clonal hematopoiesis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Prior heart attack or coronary stent procedure >180 days before baseline imaging
* Presence of either TET2 CHIP or no CHIP variants on prior sequencing

Exclusion Criteria:

* placement of a drug-eluting stent in a proximal coronary arterial segment <180 days before baseline imaging
* prior coronary artery bypass grafting
* pregnancy or breastfeeding
* history of blood malignancy or current solid-tumor malignancy
* history of organ or stem cell transplantation
* current treatment with prescription, systemic (oral, IV [intravenous], or IM [intramuscular]) steroids or anti-inflammatory/immune suppressant medical therapies (including colchicine but excluding topical therapies, UV therapy, ASA-derivative therapies, or NSAIDS) for autoimmune/inflammatory diseases, post-transplant care, asthma, or pain
* use of oral steroids or prescription oral anti-inflammatory/immune suppressant medication for >7 days within the past 1 month
* use of IV or IM steroids or IV or IM anti-inflammatory/immune suppressant medication within the past 3 months
* known allergy to dextran's and/or DTPA and/or radiometals and/or severe allergy to iodinated contrast media
* estimated glomerular filtration rate (eGFR) < 45 ml/min/1.73 m2
* contraindications to nitroglycerin known narrow angle glaucoma, or known severe aortic stenosis
* use of phosphodiesterase type 5 inhibitor AND refusal to abstain from use of these medications within the 5 days prior to scheduled CCTA scan
* significant radiation exposure (40msV) received within the past 12 months
* concurrent enrollment in another research study judged by the investigators to interfere with the current study
* known active or recurrent hepatic disease (including cirrhosis or ALT/AST levels >3 times the upper limit oof or total bilirubin >2 times the upper limits of normal)
* history or evidence of tuberculosis (TB) (active or latent) infection or risk factor for TB
* history of ongoing, chronic or recurrent infectious disease
* suspected or proven immunocompromised state
* live vaccinations within 3 months prior to randomization visit or live vaccinations planned during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Perivascular fat attenuation index (Hounsfield units) measured by coronary computed tomography angiography | 48 weeks

SECONDARY OUTCOMES:
Aortic volume with 99mTc-tilmanocept uptake (percent of aortic volume) measured by single-photon emission computed tomography | 48 weeks
TET2 variant allele fraction (proportion of mutated alleles in peripheral blood cells) ascertained by targeted genomic sequencing | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of MGH. All samples and images being analyzed by outside vendors will be de-identified